CLINICAL TRIAL: NCT03148717
Title: Preoperative vs. Postoperative Rectal Misoprostol in Cesarean Section: A Randomized, Double Blind Clinical Trial
Brief Title: Preoperative vs. Postoperative Rectal Misoprostol in Cesarean Section
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AS1380
Record Dates: First submitted 2017-04-29; First posted 2017-05-11 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Neonatal Outcome
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative (Active Comparator): Group no.1 will receive preoperative rectal 400 microgram of misoprostol (Sigma) "2 tablets" and postoperative rectal placebo"2 tablets".
  Interventions: Drug: Misoprostol; Other: Placebo
- Postoperative (Active Comparator): Group no.2 will receive preoperative rectal placebo "2 tablets" and postoperative rectal 400 microgram of misoprostol (Sigma) " 2 tablets" .
  Interventions: Drug: Misoprostol; Other: Placebo

INTERVENTIONS:
Drug: Misoprostol — Cytotec
  Other Names: Mesotac
Other: Placebo — Placebo tablet similar in shape, odour and consistency to misoprostol tablet.

SUMMARY:
This prospective double-blind placebo-controlled randomized clinical trial will be conducted at Ain-Shams University Maternity Hospital from April 2017 till December 2017. Group 1 women, candidates for cesarean section, will receive preoperative rectal 400 microgram of misoprostol, and Group 2 women will receive postoperative rectal 400 microgram of misoprostol.

2017. 120 women candidate foe elective cesarean section will receive preoperative sublingual 400 microgram of misoprostol, and another 120 women will receive postoperative sublingual 400 microgram of misoprostol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients candidate for cesarean section.
2. Full term pregnancies (GA 37- 42 Wks).
3. Age (18-40 yrs).
4. body mass index (BMI) (20-30(Kg/m2 .

Exclusion Criteia:

1. Contraindication to spinal anesthesia.
2. Blood dyscrasias.
3. Large fibroids.
4. Contraindications to prostaglandin therapy (e.g. history of severe bronchial asthma or allergy to misoprostol.
5. Emergency CS such as fetal distress
6. Extreme of BMI (<20 or >30 Kg/m2 ).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Neonatal outcome | 5 minutes
  measured by APGAR score at 5 minutes

SECONDARY OUTCOMES:
NICU admission | 24 hours
  Number of neonates admitted to NICU within 24 hours.
amount of blood loss | 24 hours
Postpartum hemorrhage | 24 hours
Need for extra uterotonics | 24 hours

OTHER OUTCOMES:
APGAR score at 1 minute | 1 minute

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt